CLINICAL TRIAL: NCT04196959
Title: An Acceptability Study to Evaluate the Adherence, Tolerance and Metabolic Control of Patients With Tyrosinaemia, When Using TYR Sphere (a Food for Special Medical Purposes (FSMP)) as Part of Dietary Management.
Brief Title: Evaluation of TYR Sphere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCT-TYRS-2019-03-04
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Tyrosinemias; Alkaptonuria; Tyrosinemia, Type I; Tyrosinemia, Type II; Tyrosinemia, Type III
Keywords: Tyrosinaemia; AKU; Food for Special Medical Purposes
MeSH Terms: conditions — Tyrosinemias; Alkaptonuria

STUDY DESIGN:
Intervention Model Description: Single group, open label.
Masking Description: Non-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients will receive TYR sphere, a Food for Special Medical Purposes, as part of thier restricted diet for 28 consecutive days.
  Interventions: Dietary Supplement: TYR sphere

INTERVENTIONS:
Dietary Supplement: TYR sphere — TYR sphere is a powdered protein substitute for patients with tyrosinaemia.

SUMMARY:
For 28 days, 20 patients with tyrosinaemia will take TYR sphere as part of the usual dietary management of their condition. Patients will record their adherence to recommended intakes each day, gastrointestinal symptoms (if any) experienced each day of weeks one and four, and the palatability of the product at the end of the trial. Metabolic control will be evaluated by dried blood spots collected during the Baseline and End of Study visits, and weekly during the 28 days of the study itself.

Trial data will be used in an application to make TYR sphere available via the NHS.

DETAILED DESCRIPTION:
TYR sphere is a glycomacropeptide (GMP) based protein substitute for patients with tyrosinaemia.

The Evaluation of TYR sphere study has been designed to generate data required by the United Kingdom's Advisory Committee on Borderline Substances (ACBS), the national regulator for Foods for Special Medical Purposes (FSMP).

The ACBS specify that before a FSMP can be routinely prescribed by the NHS, its acceptability must first be evaluated by a clinical trial in patients for whom it is ultimately designed. The ACBS define acceptability as comprising patient evaluations of the product's palatability, data on their adherence to recommended intakes and their gastrointestinal tolerance of it. TYR sphere is designed for patients of three years of age and upwards. This has informed the trial's age-related inclusion criteria.

Using a mobile phone application, or paper diary form, patients will record their intake of TYR sphere along with the recommended amount on each of the 28 study days. Gastrointestinal tolerance will be recorded each day during weeks one and four, while palatability of TYR sphere will be recorded at the end of the 28 days, or immediately on discontinuing TYR sphere if the patient stops the trial early. An evaluation of the patient's previous protein substitute and usual GI symptoms are recorded on day one, before the first intake of TYR sphere.

Metabolic control, measured via dried blood spots taken at both visits, and weekly during the 28 days study period, is another primary outcome measure alongside acceptability.

The trial's secondary endpoint is evaluations of growth. Height and weight will be recorded at the Baseline and End of Study visits.

If it is deemed appropriate by the investigator, patients may continue to take the product at the end of the Evaluation Period as part of Care After Research. This continued supply would be given free of charge by the sponsor up until the product is available via a regular prescription, having completed the registration process with the ACBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with tyrosinaemia.
* Aged ≥ 3 years.
* In the opinion of the Investigator, can comply with the study protocol and take at least one sachet of the study product per day.
* Willingly given, written, informed consent from patient or parent/guardian.
* Willingly given, written assent (if appropriate).

Exclusion Criteria:

* Individuals who are allergic to milk, fish and soya (these allergens are inherent in the study product ingredients).
* Use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the Investigator (must be recorded in patient case report form CRF).
* Women who are pregnant / breastfeeding at the start of the study or planning to become pregnant during the study period.
* Individuals who, in the opinion of the investigator, are unable to comply with the requirements of the protocol.
* Any co-morbidity, which, in the opinion of the Investigator, would preclude participation in the study.
* Patients who are currently participating in, plan to participate in, or have participated in an interventional investigational drug, food or medical device trial within 30 days prior to screening visit.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed intake of TYR sphere | Days 1 to 28
  Patient reported data on actual compared to prescribed intakes of TYR sphere
Patient record of gastrointestinal tolerance, week 1 | Days 1 - 7
  Patient reported data on any gastrointestinal symptoms experienced
Patient record of gastrointestinal tolerance, week 4 | Days 21 - 28
  Patient reported data on any gastrointestinal symptoms experienced
Patient assessment of palatability of TYR sphere | Day 28
  Patient reported data on the taste, texture, appearance, smell and ease of use of TYR sphere at the end of the trial period.
Change in metabolic control (tyrosine) over study period | One at Baseline Visit (Day 1) one per week during Evaluation Period (Days 1 - 28) and one at End of Study visit (Day 28)
  Tyrosine levels obtained from dried blood spots
Change in metabolic control (phenylalanine) over study period | One at Baseline Visit (Day 1) one per week during Evaluation Period (Days 1 - 28) and one at End of Study visit (Day 28)
  Phenylalanine levels obtained from dried blood spots

SECONDARY OUTCOMES:
Change in height | Baseline Visit (Day 1) and End of Study Visit (Day 28)
  Change in height over study period
Change in weight | Baseline Visit (Day 1) and End of Study Visit (Day 28)
  Change in weight over study period

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Anita.MacDonald@NHS.Net
Locations (2):
- United Kingdom (2):
  - National Alkaptonuria Centre, Royal Liverpool University Hospital, Liverpool, Merseyside
  - Birmingham Children's Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No